CLINICAL TRIAL: NCT00964756
Title: A Phase I Study of AD5.SSTR/TK.RGD; A Tropism Modified Adenovirus Vector for Intraperitoneal Delivery of Therapeutic Genes and Additional Capability of Noninvasive Imaging of Gene Transfer in Patients With Recurrent Ovarian and Other Selected Gynecologic Cancers (Infectivity Enhanced Adenoviral Vectors for Ovarian CA)
Brief Title: A Study of an Infectivity Enhanced Suicide Gene Expressing Adenovirus for Ovarian Cancer in Patients With Recurrent Ovarian and Other Selected Gynecologic Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ronald D. Alvarez, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F080807013 (UAB 0821); 5R01CA090547-02 (NIH); OGCA Link # 000137326 (Other: UAB); UAB 0821 (Other: UAB Department)
Record Dates: First submitted 2009-06-11; First posted 2009-08-25 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; Recurrent ovarian cancer and other gynecologic cancers
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gene therapy (Experimental)
  Interventions: Genetic: Ad5.SSTR/TK.RGD; Drug: Ganciclovir (GCV)

INTERVENTIONS:
Genetic: Ad5.SSTR/TK.RGD — Group 1 Day 1-3 IP 1 x 10 9th vp/d Group 2 Day 1-3 IP 5 x 10 10th vp/d Group 3 Day 1-3 IP 1 x 10 12th vp/d
Drug: Ganciclovir (GCV) — GVC Day 5-18 IV 5 mg/kg BID all groups

SUMMARY:
In spite of surgical and chemotherapeutic advances, long term survival for advanced and recurrent gynecologic cancers remains dismal and no curative treatment for recurrent disease exists. Novel treatment strategies are needed. This is a study to determine the maximally tolerated dose of and toxicities associated with intraperitoneal delivery of an infectivity enhanced adenovirus that expresses a suicide gene and an gene that allows imaging of gene transfer. This vector will be given in combination with intravenous ganciclovir in patients with recurrent ovarian and other gynecological cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented invasive epithelial ovarian, extraovarian, fallopian tube or endometrial carcinoma.
* Patients must have persistent or recurrent disease after standard debulking/staging surgery and conventional therapy.
* Patients must have evidence of intraabdominal disease; disease may be measurable or nonmeasurable.
* Patients must have a GOG performance status of 0, 1, or 2, and have a life expectancy of greater than 3 months.
* Patients must have adequate hematologic, renal, and hepatic function defined as:

  * WBC > 3,000 ul
  * Granulocytes > 1,500 ul
  * Platelets > 100,000
  * Creatinine clearance > 80 mg/dl or serum creatinine > 2.0
  * Serum transaminases < 2.5 x upper limits of normal
  * Normal serum bilirubin
  * PT/PTT/INR < 1.5 x institutional ULN
  * O2 saturation > or = 92 %
* Patients must be 19 years or older and must have signed informed consent

Exclusion Criteria:

* Patients with epithelial tumors of low malignant potential, stromal tumors and germ cell tumors of the ovary are ineligible to participate in the study.
* Patients with the only site of disease located beyond the abdominal cavity are ineligible to participate in the study.
* Patients who are pregnant or lactating are ineligible to participate in the study.
* Patients with a GOG performance status of 3 or 4 are ineligible to participate in the study.
* Patients with active heart disease (characterized by angina, unstable arrhythmia, congestive heart failure or EF < 55%, pulmonary hyper- tension, active or chronic debilitating pulmonary disease(i.e., active pneumonia, severe COPD, pulmonary edema, O2 saturation < 92%), or coagulation disorders (i.e. bleeding disorders, or on therapeutic anti- coagulants)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Evaluation for toxicity | 2 years

SECONDARY OUTCOMES:
Molecular Studies for evaluation of gene transfer and generation of wild type adenovirus, viral shedding and clinical efficacy | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Alvarez, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] Kim KH, Dmitriev I, O'Malley JP, Wang M, Saddekni S, You Z, Preuss MA, Harris RD, Aurigemma R, Siegal GP, Zinn KR, Curiel DT, Alvarez RD. A phase I clinical trial of Ad5.SSTR/TK.RGD, a novel infectivity-enhanced bicistronic adenovirus, in patients with recurrent gynecologic cancer. Clin Cancer Res. 2012 Jun 15;18(12):3440-51. doi: 10.1158/1078-0432.CCR-11-2852. Epub 2012 Apr 17. PMID 22510347